CLINICAL TRIAL: NCT01571037
Title: Inhaled Milrinone Use in Patients Receiving HeartMate II LVAD: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0195-11-FB
Record Dates: First submitted 2011-05-06; First posted 2012-04-04 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: End Stage Heart Disease; Right Ventricular Dysfunction
Keywords: mechanical circulatory assist device
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Inhalation; Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inhaled nebulized Milrinone (Other): Drug: Inhaled, nebulized, Milrinone
  1 mg/ml milrinone (dissolved in dextrose) and diluted in 0.9% normal saline in a 1:1 ratio to final drug concentration of 0.5mg/ml will be delivered via an IV pump at a fixed dose of 12 ml/hour which will run into a vibrating mesh nebulizer reservoir, connected to the mechanical ventilator circuit. Inhaled milrinone will begin at time of resumption of mechanical ventilation when initiating wean from cardiopulmonary bypass after LVAD implantation in the operating room, and run continuously for a total maximum duration of 24 hours OR until the patient is extubated whichever occurs first. Plasma milrinone levels will be assessed to determine if systemic milrinone absorption occurs after prolonged milrinone inhalation.
  Interventions: Drug: Inhaled, nebulized, Milrinone; Drug: inhaled nebulized milrinone

INTERVENTIONS:
Drug: Inhaled, nebulized, Milrinone — 1 mg/ml milrinone (dissolved in dextrose) and diluted in 0.9% normal saline in a 1:1 ratio to final drug concentration of 0.5mg/ml will be delivered via an IV pump at a fixed dose of 12 ml/hour which will run into a vibrating mesh nebulizer reservoir, connected to the mechanical ventilator circuit. Inhaled milrinone will begin at time of resumption of mechanical ventilation when initiating wean from cardiopulmonary bypass after LVAD implantation in the operating room, and run continuously for a total maximum duration of 24 hours OR until the patient is extubated whichever occurs first. Plasma milrinone levels will be assessed to determine if systemic milrinone absorption occurs after prolonged milrinone inhalation.
  Other Names: Primacor
Drug: inhaled nebulized milrinone — 0.5 mg/ml inhaled nebulized milrinone deliver at 12 ml/hr continuously until either 24 hours or extubated.
  Other Names: Primacor

SUMMARY:
Right ventricular (RV) failure occurs in an estimated 5-41% of cases involving left ventricular assist device (LVAD) implantation and has been shown to adversely affect peri-operative morbidity and mortality. Current therapies to improve RV dysfunction pre and post-operatively are limited. Inhaled milrinone has been shown in several small human studies to be safely tolerated and provide favorable effects on pulmonary hemodynamics.

Study Hypothesis: Delivery of inhaled milrinone, a phosphodiesterase III inhibitor, may provide pulmonary artery vasodilation and therefore improved RV function in patients with end stage heart failure receiving HeartMate II LVAD as a bridge to cardiac transplantation or as destination therapy.

Specifically, we aim to:

* demonstrate safety of inhaled milrinone in this patient cohort
* demonstrate efficacy of inhaled milrinone in this patient cohort

DETAILED DESCRIPTION:
Right ventricular (RV) failure occurs in an estimated 5-41% of cases involving left ventricular assist device (LVAD) implantation and has been shown to adversely affect peri-operative morbidity and mortality. Current therapies to improve RV dysfunction pre and post-operatively are limited. Inhaled milrinone has been shown in several small human studies to be safely tolerated and provide favorable effects on pulmonary hemodynamics.

Study Hypothesis: Delivery of inhaled milrinone, a phosphodiesterase III inhibitor, may provide pulmonary artery vasodilation and therefore improved RV function in patients with end stage heart failure receiving HeartMate II LVAD as a bridge to cardiac transplantation or as destination therapy.

Specifically, the aims are:

demonstrate safety of inhaled milrinone in this patient cohort demonstrate efficacy of inhaled milrinone in this patient cohort

ELIGIBILITY:
Inclusion Criteria:

1. For BTT candidates:

   * Must be an approved candidate for heart transplantation according to institutional policy
2. For DT candidates:

   * Patients with New York Heart Association (NYHA) class IV symptoms that have failed to respond to maximal medical therapy including beta blocker and angiotensin converting enzyme inhibitors if tolerated for at least 45 of 60 days, OR dependence on continuous inotropic therapy for 14 days OR dependence on intra-aortic balloon pump (IABP) for 7 days
   * Left ventricular ejection fraction (LVEF) < 25%
   * Patients with functional limitations on cardiopulmonary stress testing with a peak oxygen consumption of ≤ 14 ml/kg/min unless balloon pump or inotrope dependent or physically unable to perform the test.
   * Patients not deemed to be a heart transplant candidate after evaluation
   * Must have mean PAP > 25 mmHg by pulmonary catheter indices pre-operatively (within 72 hrs) and/or a PVR > 3 Woods units (WU).
   * Age ≥ 19 years old (in the state of Nebraska, an individual must be ≥ 19 years old to legally provide consent as compared to age ≥ 18 in most other states)
   * Signed informed consent

Exclusion Criteria:

* Age < 19 years old
* Pregnancy or current breast feeding
* Undergoing cardiac transplantation without implantation of mechanical assist device
* Documented medical allergy to milrinone
* Failure to meet inclusion criteria for LVAD implantation for BTT or DT indications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04-05 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2014-02-21 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of Arrhythmias, Hypotension and Hypersensitivity Reaction | 12 and 24 hours
  1. Arrhythmias:
     * Atrial
     * Ventricular
  2. 'Sustained' hypotension
  3. Hypersensitivity reaction to milrinone

SECONDARY OUTCOMES:
Efficacy - Hemodynamic | 30, 60 minutes, then every 4 hours thereafter
  Invasive Hemodynamic pulmonary catheter:
  * PAS, PAD, mPAP, RA pressures, PCWP, CI, RVSWi (calculated), TPG, PVR, and SvO2
Efficacy - Echocardiographic | Pre-op Echocardiography, intraoperative TEE (before and after inhaled milrinone) and postoperative Echocardiography within 48 hours of milrinone initiation
  Echocardiographic
  * RV dimensions
  * RV systolic functional assessment
  * Tricuspid valve regurgitation
  * Pulmonary Vascular resistance

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Haglund, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States